CLINICAL TRIAL: NCT04283175
Title: Validation Study of Posturology Platforms and Exploratory Study for Evaluating Postural Control of Hemiparetic and Neuro-muscular Patients
Brief Title: Validation Study of Posturology Platforms for Evaluating Postural Control of Hemiparetic and Neuro-muscular Patients
Acronym: KPLATES
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Motion analysis laboratory, Garches (Unknown); Fondation de Garches (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP19974; 2019-A02392-55 (Registry Identifier: IDRCB)
Record Dates: First submitted 2020-02-20; First posted 2020-02-25 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Neuromuscular Diseases; Hemiparesis; Charcot-Marie-Tooth Disease
Keywords: Neuromuscular Diseases; Charcot-Marie-Tooth Disease; Hemiparesis
MeSH Terms: conditions — Neuromuscular Diseases; Paresis; Charcot-Marie-Tooth Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Neuromuscular disease (MNM) subjects (Charcot Marie Tooth disease, CMT)
  Interventions: Other: Posturological examination on KPlates and AMTI platforms; Other: Berg Balance Scale (BBS)
- Hemiparetic subjects
  Interventions: Other: Posturological examination on KPlates and AMTI platforms; Other: Berg Balance Scale (BBS)
- Healthy subjects
  Interventions: Other: Posturological examination on KPlates and AMTI platforms

INTERVENTIONS:
Other: Posturological examination on KPlates and AMTI platforms — By an unique evaluator
Other: Berg Balance Scale (BBS) — Falls and fera of falling, motor and sensory impairments
  Groups: Hemiparetic subjects; Neuromuscular disease (MNM) subjects (Charcot Marie Tooth disease, CMT)

SUMMARY:
The instrumental evaluation of standing postural control by posturographic analysis supplements the clinical evaluation and, as such, is recommended by the French National Authority for Health (HAS 2007). The quantitative data obtained after a standardized postural examination appear relevant for the longitudinal follow-up of neuromuscular patients and hemiparetic patients. Neuro muscular (NM) diseases are progressive, these instrumental evaluations can highlight a deterioration or stabilization of postural control possibly not observable with the scores on clinical scales.

The K-Force Plates, recently developed appear to be an interesting alternative to the stabilometry platforms currently used. Static and dynamic conditions in upright position are tested. Moreover, posturologic, kinematics data and clinical scores are correlated to increase understanding of strategies during postural control tasks in patients with stroke and in patients with NM disorders.

DETAILED DESCRIPTION:
To date, no clinical validation study of these K-Force Plates force platforms has been proposed. The investigator hypothesize that the data obtained by the Plates are comparable to the measurements made by the reference tool, the AMTI platforms during a static and dynamic posturographic examination in MNM, hemiparetic and healthy subjects. The strategies of the patients (stroke and NM) during the dynamic task are also explored with kinematic analysis in correlation with data from force platforms and clinical scores.

ELIGIBILITY:
"Eligible couples must present all the following criteria :

* Signing of the informed consent form
* Men and women aged from 18
* Single stroke hemiparetic patient, or patient with neuro-muscular disease, or healthy subject free of neurological disorder and other disease
* Patient able to stand alone at least 30 seconds without technical assistance (multiple repetitions)

To be included, patient should not present any of the following criteria :

* Bilateral brain injury, cerebellar syndrome
* Other disease or defect that may interfere with the study such as visual, vestibular or other related uncontrolled medical condition
* Major cognitive impairment that does not allow evaluation
* Pregnant women, breastfeeding
* Non affiliated to a social security scheme"

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Single stroke hemiparetic patient, or patient with neuro-muscular disease, or healthy subject free of neurological disorder and other disease.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Evaluate the concurrent validity of K-Force Plates (K-Invent) force platforms in comparison with reference platforms (AMTI) for posturological examination in static and dynamic conditions of MNM subjects (CMT), hemiparetic subjects and healthy subjects. | Day 0
  Intraclass correlation coefficient (ICC) of the mean velocity of the pressure center (CP) with the both platforms during the posturological examination. The average of 3 tests carried out will be taken

SECONDARY OUTCOMES:
Evaluate convergent validity with the reference scale for the assessment of equilibrium disorders | Day 0
  Berg's equilibrium rating scale (0-56) ( score at 0: worse outcome)
Compare the posturology and kinematics between stroke and healthy subjects and between NM and healthy subjects | Day 0
  Explore the relations between the posturology, kinematics and clinical parameters in stroke population and in NM population.

CONTACTS AND LOCATIONS:
Overall Officials: Celine Bonnyaud, PhD, Principal Investigator — Laboratoire d'analyse du mouvement, Hopital Raymond Poincaré, APHP
Locations (1):
- Laboratoire d'analyse du mouvement, Hopital Raymond Poincaré, APHP, Garches, France